CLINICAL TRIAL: NCT04826094
Title: A Randomized, Double-Blind Phase 1 Trial to Evaluate the Safety and Immunogenicity of Priming With Env-C Plasmid DNA Vaccine Alone, With Different Adjuvants, or With an Adjuvanted HIV Env gp145 C.6980 Protein Vaccine and Boosting With the Adjuvanted HIV Env gp145 C.6980 Protein Vaccine With or Without the Env-C Plasmid DNA Vaccine in Healthy HIV Uninfected Adults in Kenya
Brief Title: A Study to Assess the Safety and Immune Response to Env-C DNA and Protein Vaccines in Kenya
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); US Military HIV Research Program (Network); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RV460; 38608 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2023-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group 1: Vaccine (Experimental): 3 doses of prime vaccination at weeks 0, 4, 12 followed by 3 doses of boost vaccination at weeks 20, 32, 56
  Interventions: Biological: Env-C Plasmid DNA; Biological: HIV Env gp145 C.6980 protein; Drug: Rehydragel®; Drug: Placebo (IM)
- Group 2: Vaccine (Experimental): 3 doses of prime vaccination at weeks 0, 4, 12 followed by 3 doses of boost vaccination at weeks 20, 32, 56
  Interventions: Biological: Env-C Plasmid DNA; Biological: HIV Env gp145 C.6980 protein; Drug: Rehydragel®; Biological: ALF43; Drug: Placebo (IM)
- Group 3: Vaccine (Experimental): 3 doses of prime vaccination at weeks 0, 4, 12 followed by 3 doses of boost vaccination at weeks 20, 32, 56
  Interventions: Biological: Env-C Plasmid DNA; Biological: HIV Env gp145 C.6980 protein; Drug: Rehydragel®; Biological: dmLT; Drug: Placebo (IM); Drug: Placebo (TCl)
- Group 4: Vaccine (Experimental): 3 doses of prime vaccination at weeks 0, 4, 12 followed by 3 doses of boost vaccination at weeks 20, 32, 56
  Interventions: Biological: Env-C Plasmid DNA; Biological: HIV Env gp145 C.6980 protein; Drug: Rehydragel®; Biological: ALF43; Biological: dmLT; Drug: Placebo (IM); Drug: Placebo (TCl)
- Group 5: Vaccine (Experimental): 3 doses of prime vaccination at weeks 0, 4, 12 followed by 3 doses of boost vaccination at weeks 20, 32, 56
  Interventions: Biological: Env-C Plasmid DNA; Biological: HIV Env gp145 C.6980 protein; Drug: Rehydragel®; Biological: ALF43; Drug: Placebo (IM)
- Group 6: Vaccine (Experimental): 3 doses of prime vaccination at weeks 0, 4, 12 followed by 3 doses of boost vaccination at weeks 20, 32, 56
  Interventions: Biological: Env-C Plasmid DNA; Biological: HIV Env gp145 C.6980 protein; Drug: Rehydragel®; Biological: ALF43; Drug: Placebo (IM)
- Group 7: Vaccine (Experimental): 3 doses of prime vaccination at weeks 0, 4, 12 followed by 3 doses of boost vaccination at weeks 20, 32, 56
  Interventions: Biological: Env-C Plasmid DNA; Biological: HIV Env gp145 C.6980 protein; Drug: Rehydragel®; Biological: ALF43; Drug: Placebo (IM)
- Pooled Placebo (Placebo Comparator): Pooled placebo arm.
  Interventions: Drug: Placebo (TCl)

INTERVENTIONS:
Biological: Env-C Plasmid DNA — 2 mg per dose. Administered by intramuscular injection.
  Arms: Group 1: Vaccine; Group 2: Vaccine; Group 3: Vaccine; Group 4: Vaccine; Group 5: Vaccine; Group 6: Vaccine; Group 7: Vaccine
Biological: HIV Env gp145 C.6980 protein — 100 µg per dose. Administered by intramuscular injection.
  Arms: Group 1: Vaccine; Group 2: Vaccine; Group 3: Vaccine; Group 4: Vaccine; Group 5: Vaccine; Group 6: Vaccine; Group 7: Vaccine
Drug: Rehydragel® — Adjuvant. Aluminum hydroxide fluid gel. 500 µg per dose. Administered by intramuscular injection.
  Arms: Group 1: Vaccine; Group 2: Vaccine; Group 3: Vaccine; Group 4: Vaccine; Group 5: Vaccine; Group 6: Vaccine; Group 7: Vaccine
Biological: ALF43 — Adjuvant. Army Liposome Formulation-43% Cholesterol. 200 µg per dose. Administered by intramuscular injection.
  Arms: Group 2: Vaccine; Group 4: Vaccine; Group 5: Vaccine; Group 6: Vaccine; Group 7: Vaccine
Biological: dmLT — Adjuvant. Recombinant double mutant Escherichia coli heat labile toxin. 50 µg per dose. Transcutaneous application (needle-free skin patch). 1 mL diluted dmLT added to gauze pad at site of injection.
  Arms: Group 3: Vaccine; Group 4: Vaccine
Drug: Placebo (IM) — 0.9% sodium chloride (sterile saline). Administered by intramuscular injection.
  Arms: Group 1: Vaccine; Group 2: Vaccine; Group 3: Vaccine; Group 4: Vaccine; Group 5: Vaccine; Group 6: Vaccine; Group 7: Vaccine
Drug: Placebo (TCl) — Transcutaneous application (needle-free skin patch). 0.9% sodium chloride (sterile saline) added to gauze pad at site of injection.
  Arms: Group 3: Vaccine; Group 4: Vaccine; Pooled Placebo

SUMMARY:
This is a study of HIV vaccines. A vaccine is a medical product given to prevent certain diseases. The vaccine may educate the body to form a defensive response to try to prevent the disease from the beginning, or preventing it from taking hold of the body. This defensive response is called the immune response. The experimental vaccines in this study are Env-C Plasmid DNA and HIV Env gp145 C690 protein, given with different adjuvants. An adjuvant is a substance added to vaccines that can help make the vaccine more effective by improving the immune response, or by causing the immune response to last longer than it would without the adjuvant. The adjuvants are mixed with the vaccines and injected into muscle or placed on top of the skin. The HIV vaccines contain a piece of genetic material or a protein copied drom the HIV virus cover (Env), but they do not contain the virus itself. The vaccines cannot cause HIV infection or Acquired Immune Deficiency Syndrome (AIDS).

The purpose of this study is to find out if the study vaccines with adjuvants cause side effects and are tolerable, whether humans respond (develop immune responses) to the vaccines, and how ling the effects of the study vaccines last. The study will also compare the effects of the study vaccines with adjuvants and adjuvant patch to those of placebo injections and placebo patch. The placebo will consist of saline (sterile saltwater) and will look like study vaccines, be given in the same way, but will have no active vaccine or adjuvant in it. A total of 126 participants will take part in the study and each will have up to 26 clinic visits and will be followed-up for a total of 108 weeks.

DETAILED DESCRIPTION:
Antibodies are the most commonly recognized correlate of vaccine protection from infection; however the possible protective HIV antibody levels, which were induced by the modestly protective RV144 vaccine regimen with alum, rapidly decayed. Potentially, a novel, highly selective adjuvant combined with the correctly sequenced HIV antigen could slow antibody decay, increase antibody magnitude and induce antibodies of appropriate functional response.

RV460 is an exploratory study that will assess the safety, tolerability, and immunogenicity of a vaccine regimen consisting of priming with an Env-C Plasmid DNA vaccine (with or without novel adjuvants) when given with or without adjuvanted HIV Env gp145 C.6980 protein vaccine and boosting with adjuvanted gp145 C.6980 protein with or without the gp120 DNA vaccine. The study will be carried out in Kericho, Kenya. 126 healthy adults will ben enrolled. Participants will be randomized into one of seven groups which have 15/3 vaccine/placebo recipients per group. Each participant will receive six injections (prim at week 0, 4, 12; boost at week 20, 32 and 56) and will be followed-up for a total of 108 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male and female participant aged 18 to 40 years and available for 26 months.
* Must be at low risk for HIV infection per investigator assessment and using the study risk assessment tool.
* Must be able to understand and complete the informed consent process.
* Must be capable of reading English or Kiswahili.
* Must agree to a home visit.
* Must complete a Test of Understanding (TOU) before enrollment. Must answer 9 out of 10 questions correctly with a maximum of three attempts.
* Must be in good general health without a clinically significant medical history.
* HIV-uninfected per diagnostic algorithm within 45 days of enrollment.
* Laboratory values:

  * Hemoglobin

    * 12.5-18.1 g/dL men
    * 11.0-16.1 g/dL women
  * White Cell Count

    * 2.7-7.7 x 10³ cells/µL men
    * 3.0-9.1 x 10³ cells/µL women
  * Platelets:

    * 125-370 10³ cells/µL men
    * 125-444 10³ cells/µL women
  * ALT and AST: ≤1.25 institutional upper limit of the reference range
  * Creatinine: ≤1.25 institutional upper limit of the reference range
  * Urinalysis: (dipstick) for blood and protein less than 1+ and negative glucose Female-Specific Criteria
* Negative urine pregnancy test for women at screening, the day of each vaccination, and before any invasive procedure.
* Already using and commits to continued use of an adequate birth control method for 45 days before to the first vaccination/placebo vaccination, and for at least 90 days after the final vaccine/placebo vaccination. Adequate birth control is defined as follows: Contraceptive medications delivered orally, intramuscularly, vaginally, or implanted, underneath the skin, surgical methods (hysterectomy or bilateral tubal ligation), condoms with spermicide, diaphragms, intrauterine device (IUD), vasectomy in a monogamous partner, or abstinence.

Lymph Node Biopsy Inclusion Criteria

* Body mass index (BMI) <35
* Platelets >150,000
* International normalized ration (INR) <1.2
* Verbal report of no NSAIDS/aspirin for 7 days prior.
* Negative pregnancy test for participants born female.

Exclusion Criteria:

A history of:

* Three or more sexual partners in the previous 24 weeks.
* Commercial sex work.
* Non-adherence to condom use in the absence of a long-term monogamous relationship.
* Intravenous drug use in the previous year.
* A sexually transmitted infection in the previous 24 weeks.
* Asplenia: any condition resulting in the absence of a functional spleen.
* Bleeding disorder diagnosed by a medical doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions).
* Breastfeeding or pregnant (positive pregnancy test) women or planning to become pregnant during the window between study enrollment and three months after the last vaccination visit.
* Any past, ongoing, or in remission history of treated or untreated autoimmune disease.
* Has known active Hepatitis B virus infection (or positive HBsAg).
* Has known active Hepatitis C infection.
* History of anaphylaxis or other serious adverse reaction to vaccines or allergies or reactions likely to be exacerbated by any component of the vaccine and placebo, including antibiotics or excipients.
* Absolute Neutrophil Count (ANC) <1.0 x 10³ cells/µL.
* Participant has received any of the following substances:

  * Chronic use of therapies that may modify immune response, such as intravenous (IV) immune globulin and systemic corticosteroids (in doses of >20 mg/day prednisone equivalent for periods exceeding 10 days).
  * The following exceptions are permitted and will not exclude study participation:

    * Use of corticosteroid nasal spray for rhinitis;
    * Topical corticosteroids for an acute uncomplicated dermatitis; or
    * A short course (10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on investigator clinical judgment) at least 2 weeks before enrollment.
* Blood products within 120 days before HIV screening.
* Immunoglobulins within 30 days before HIV screening.
* Any experimental vaccine containing an adjuvant other than aluminum of an adjuvant not approved by the FDA or European Medicines Agency (EMA) as part of a licensed vaccine.
* CERVARIX vaccine against HPV (containing AS04)
* Receipt of any investigational HIV vaccine, investigational research agents or vaccine within 30 days before enrollment.
* Anti-tuberculosis prophylaxis or therapy during the past 90 days before enrollment.
* Any psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contraindication to protocol compliance or impairs a participant's ability to give informed consent.
* Major psychiatric illness and or substance abuse problems during the past 12 months that, in the opinion of the investigator, would preclude participation.
* History of atopy or significant skin conditions.
* Study site employees who are involved in the protocol and or may have direct access to the study-related area.

Lymph Node Biopsy Exclusion Criteria

* History of keloid formation.
* History of an inguinal hernia, inguinal canal cryptorchidism, varicocele, hydrocele.
* History of inguinal excisional lymph node biopsy.

Final evaluation of eligibility is based on the medical judgment of the investigator. The Protocol Safety Review Team will also remain available to the investigator for consultation if desired.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josphat Kosgei, MBChB, MSc, Principal Investigator — Kenya Medical Research Institute/US Medical Research Directorate-Africa; Christina Polyak, MD, Study Chair — U.S. Military HIV Research Program (MHRP)/Walter Reed Army Institute of Research (WRAIR); Sandhya Vasan, MD, Study Chair — U.S. Military HIV Research Program (MHRP)/Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Kenya Medical Research Institute/Walter Reed Project, Clinical Research Centre, Off Hospital Road, Kericho, Kenya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: See protocol for screening details.
Period: Overall Study
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Pooled Placebo
Started | 17 | 16 | 17 | 16 | 16 | 18 | 17 | 26
Completed | 13 | 14 | 15 | 15 | 13 | 12 | 14 | 20
Not Completed | 4 | 2 | 2 | 1 | 3 | 6 | 3 | 6
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 1 | 3 | 1 | 1
Not completed — Participant withdrew consent | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Not completed — Non-adherence (protocol deviation) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawn by Investigator | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other: Moved from area | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other: Declined | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other: Vaccine not administered | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Pooled Placebo | Total
Number analyzed (Participants) | 17 | 16 | 17 | 16 | 16 | 18 | 17 | 26 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All Randomized Participants
  years
    Age Years | 26.4 (3.7) | 26.6 (5.3) | 29.0 (4.5) | 27.2 (5.9) | 29.2 (5.0) | 28.8 (5.2) | 28.7 (3.9) | 28.7 (6.0) | 28.1 (5.0)
Age, Customized [Count of Participants; unit: Participants]
  18-25 | 8 | 8 | 4 | 8 | 3 | 5 | 4 | 9 | 49
  26-30 | 6 | 3 | 6 | 3 | 8 | 4 | 9 | 6 | 45
  31-35 | 3 | 4 | 6 | 2 | 2 | 8 | 3 | 8 | 36
  36-40 | 0 | 1 | 1 | 3 | 3 | 1 | 1 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 13 | 9 | 8 | 11 | 12 | 15 | 86
  Male | 7 | 8 | 4 | 7 | 8 | 7 | 5 | 11 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 16 | 17 | 16 | 16 | 18 | 17 | 26 | 143
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 17 | 16 | 17 | 16 | 16 | 18 | 17 | 26 | 143
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.05 (5.13) | 22.49 (4.73) | 23.95 (3.84) | 21.87 (2.92) | 21.31 (3.30) | 22.00 (3.09) | 22.65 (3.76) | 24.37 (5.27) | 22.95 (4.23)
Tribe [Count of Participants; unit: Participants]
  Kalenjin | 12 | 15 | 16 | 15 | 11 | 17 | 15 | 20 | 121
  Kisii | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 6
  Luhya | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 6
  Luo | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 6
  Kikuyu | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Refuse to answer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Marital Status [Count of Participants; unit: Participants]
  Single, never married | 6 | 8 | 4 | 5 | 5 | 8 | 6 | 11 | 53
  Married or living as a couple | 11 | 8 | 12 | 10 | 10 | 8 | 10 | 15 | 84
  Divorced / Separated | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Widowed | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Married but living apart | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Level of Education [Count of Participants; unit: Participants]
  No formal education | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Primary school not completed | 2 | 6 | 6 | 4 | 2 | 5 | 7 | 11 | 43
  Primary school completed | 5 | 4 | 4 | 7 | 7 | 3 | 5 | 2 | 37
  Secondary school not completed | 2 | 0 | 4 | 2 | 3 | 2 | 0 | 1 | 14
  Secondary school completed | 3 | 5 | 0 | 1 | 1 | 4 | 3 | 3 | 20
  College/university | 5 | 1 | 3 | 2 | 3 | 3 | 2 | 9 | 28
  Advanced degree | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Primary Occupation [Count of Participants; unit: Participants]
  Student | 2 | 2 | 2 | 2 | 3 | 3 | 0 | 7 | 21
  Housewife | 2 | 1 | 1 | 2 | 2 | 0 | 0 | 2 | 10
  Personal or domestic services | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Unskilled laborer | 4 | 5 | 2 | 4 | 2 | 5 | 5 | 2 | 29
  Farmer | 2 | 5 | 11 | 6 | 6 | 7 | 6 | 10 | 53
  Entertainment/Services/Hospitality | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Skilled trade (tailor, hairdresser, etc.) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4
  Professional/managerial | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Commerce/business | 4 | 2 | 0 | 2 | 1 | 0 | 3 | 4 | 16
  Sex worker | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fisher/Fish trader | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Truck driver | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Military officer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Military enlisted | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Refuse to answer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Solicited Local Events Post Vaccination 1 by Priming Dose Group (Outcome 1)
Description: Incidence (number and percentage of participants) of local reactogenicity events post dose 1 by symptom, maximum severity, and priming dose group
Time Frame: Day 1-Day 7 Post Vaccination 1
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Priming Dose Group 1: Prime of Env-C Plasmid DNA Alone: Priming Dose Group 1: Prime of Env-C Plasmid DNA alone
- Priming Dose Group 2: Prime of Env-C Plasmid DNA / dmLT: Priming Dose Group 2: Prime of Env-C Plasmid DNA / dmLT
- Priming Dose Group 3: Prime of Env-C Plasmid DNA / ALF43: Priming Dose Group 3: Prime of Env-C Plasmid DNA / ALF43
- Priming Dose Group 4: Prime of Env-C Plasmid DNA / ALF43 / HIV Env gp145 C.6980 Protein: Priming Dose Group 4: Prime of Env-C Plasmid DNA / ALF43 / HIV Env gp145 C.6980 protein
- Pooled Placebo: Pooled Placebo
- All Participants Receiving Env-C Plasmid DNA: All Participants Receiving Env-C Plasmid DNA
Arm/Group | Priming Dose Group 1: Prime of Env-C Plasmid DNA Alone | Priming Dose Group 2: Prime of Env-C Plasmid DNA / dmLT | Priming Dose Group 3: Prime of Env-C Plasmid DNA / ALF43 | Priming Dose Group 4: Prime of Env-C Plasmid DNA / ALF43 / HIV Env gp145 C.6980 Protein | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 33 | 32 | 33 | 16 | 23 | 114
Participants
  Any Solicited Local Reactogenicity Event: None | 23 | 27 | 25 | 10 | 20 | 85
  Any Solicited Local Reactogenicity Event: Mild (Grade 1) | 8 | 4 | 8 | 4 | 3 | 24
  Any Solicited Local Reactogenicity Event: Moderate (Grade 2) | 2 | 1 | 0 | 2 | 0 | 5
  Any Solicited Local Reactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Local Reactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: None | 27 | 28 | 26 | 12 | 20 | 93
  Pain/Tenderness: Mild (Grade 1) | 5 | 3 | 7 | 2 | 3 | 17
  Pain/Tenderness: Moderate (Grade 2) | 1 | 1 | 0 | 2 | 0 | 4
  Pain/Tenderness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Itching: None | 29 | 30 | 32 | 14 | 23 | 105
  Itching: Mild (Grade 1) | 3 | 2 | 1 | 2 | 0 | 8
  Itching: Moderate (Grade 2) | 1 | 0 | 0 | 0 | 0 | 1
  Itching: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Itching: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: None | 28 | 32 | 33 | 14 | 22 | 107
  Warmth: Mild (Grade 1) | 5 | 0 | 0 | 2 | 1 | 7
  Warmth: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: None | 33 | 31 | 32 | 15 | 23 | 111
  Swelling/Induration: Mild (Grade 1) | 0 | 1 | 1 | 1 | 0 | 3
  Swelling/Induration: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: None | 32 | 32 | 31 | 15 | 23 | 110
  Redness/Erythema: Mild (Grade 1) | 1 | 0 | 2 | 1 | 0 | 4
  Redness/Erythema: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: None | 33 | 30 | 33 | 15 | 23 | 111
  Hardness: Mild (Grade 1) | 0 | 2 | 0 | 0 | 0 | 2
  Hardness: Moderate (Grade 2) | 0 | 0 | 0 | 1 | 0 | 1
  Hardness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Solicited Local Events Post Vaccination 2 by Priming Dose Group (Outcome 2)
Description: Incidence (number and percentage of participants) of local reactogenicity events post dose 2 by symptom, maximum severity, and priming dose group
Time Frame: Day 1-Day 7 Post Vaccination 2
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Priming Dose Group 1: Prime of Env-C Plasmid DNA Alone | Priming Dose Group 2: Prime of Env-C Plasmid DNA / dmLT | Priming Dose Group 3: Prime of Env-C Plasmid DNA / ALF43 | Priming Dose Group 4: Prime of Env-C Plasmid DNA / ALF43 / HIV Env gp145 C.6980 Protein | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 30 | 25 | 31 | 15 | 20 | 101
Participants
  Any Solicited Local Reactogenicity Event: None | 26 | 19 | 28 | 11 | 18 | 84
  Any Solicited Local Reactogenicity Event: Mild (Grade 1) | 4 | 6 | 3 | 4 | 2 | 17
  Any Solicited Local Reactogenicity Event: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Local Reactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Local Reactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: None | 27 | 19 | 28 | 11 | 19 | 85
  Pain/Tenderness: Mild (Grade 1) | 3 | 6 | 3 | 4 | 1 | 16
  Pain/Tenderness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Itching: None | 29 | 23 | 28 | 13 | 20 | 93
  Itching: Mild (Grade 1) | 1 | 2 | 3 | 2 | 0 | 8
  Itching: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Itching: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Itching: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: None | 30 | 24 | 31 | 14 | 19 | 99
  Warmth: Mild (Grade 1) | 0 | 1 | 0 | 1 | 1 | 2
  Warmth: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: None | 30 | 24 | 31 | 13 | 20 | 98
  Swelling/Induration: Mild (Grade 1) | 0 | 1 | 0 | 2 | 0 | 3
  Swelling/Induration: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: None | 30 | 25 | 31 | 14 | 20 | 100
  Redness/Erythema: Mild (Grade 1) | 0 | 0 | 0 | 1 | 0 | 1
  Redness/Erythema: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: None | 30 | 25 | 31 | 14 | 20 | 100
  Hardness: Mild (Grade 1) | 0 | 0 | 0 | 1 | 0 | 1
  Hardness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Solicited Local Events Post Vaccination 3 by Priming Dose Group (Outcome 3)
Description: Incidence (number and percentage of participants) of local reactogenicity events post dose 3 by symptom, maximum severity, and vaccination group.
Time Frame: Day 1-Day 7 Post Vaccination 3
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Priming Dose Group 1: Prime of Env-C Plasmid DNA Alone | Priming Dose Group 2: Prime of Env-C Plasmid DNA / dmLT | Priming Dose Group 3: Prime of Env-C Plasmid DNA / ALF43 | Priming Dose Group 4: Prime of Env-C Plasmid DNA / ALF43 / HIV Env gp145 C.6980 Protein | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 30 | 24 | 30 | 14 | 20 | 98
Participants
  Any Solicited Local Reactogenicity Event: None | 25 | 23 | 26 | 14 | 19 | 88
  Any Solicited Local Reactogenicity Event: Mild (Grade 1) | 5 | 1 | 4 | 0 | 1 | 10
  Any Solicited Local Reactogenicity Event: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Local Reactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Local Reactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: None | 25 | 23 | 28 | 14 | 19 | 90
  Pain/Tenderness: Mild (Grade 1) | 5 | 1 | 2 | 0 | 1 | 8
  Pain/Tenderness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Itching: None | 28 | 24 | 30 | 14 | 20 | 96
  Itching: Mild (Grade 1) | 2 | 0 | 0 | 0 | 0 | 2
  Itching: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Itching: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Itching: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: None | 29 | 24 | 29 | 14 | 20 | 96
  Warmth: Mild (Grade 1) | 1 | 0 | 1 | 0 | 0 | 2
  Warmth: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: None | 30 | 24 | 29 | 14 | 20 | 97
  Swelling/Induration: Mild (Grade 1) | 0 | 0 | 1 | 0 | 0 | 1
  Swelling/Induration: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: None | 30 | 24 | 29 | 14 | 20 | 97
  Redness/Erythema: Mild (Grade 1) | 0 | 0 | 1 | 0 | 0 | 1
  Redness/Erythema: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: None | 30 | 24 | 30 | 14 | 20 | 98
  Hardness: Mild (Grade 1) | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Solicited Local Events Post Vaccination 4 by Vaccination Group (Outcome 4)
Description: Incidence (number and percentage of participants) of local reactogenicity events post dose 4 by symptom, maximum severity, and vaccination group
Time Frame: Day 1-Day 7 Post Vaccination 4
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel®: Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 protein / Rehydragel®
- Group 2: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel®/ ALF43: Group 2: Env-C Plasmid DNA + HIV Env gp145 C.6980 protein / Rehydragel®/ ALF43
- Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel: Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 protein / Rehydragel
- Group 4: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43: Group 4: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 protein / Rehydragel® / ALF43
- Group 5: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel®: Group 5: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 protein / Rehydragel®
- Group 6: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43: Group 6: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 protein / Rehydragel® / ALF43
- Group 7:: Group 7: Env-C Plasmid DNA / HIV Env gp145 C.6980 protein / ALF43 + Env-C Plasmid DNA / HIV Env gp145 C.6980 protein / ALF43 / Rehydragel®
Arm/Group | Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 2: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel®/ ALF43 | Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel | Group 4: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 5: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 6: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 7: | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 15 | 14 | 16 | 14 | 15 | 15 | 15 | 20 | 104
Participants
  Any Solicited Local Reactogenicity Event: None | 8 | 12 | 9 | 9 | 12 | 14 | 15 | 18 | 79
  Any Solicited Local Reactogenicity Event: Mild (Grade 1) | 6 | 2 | 7 | 4 | 3 | 1 | 0 | 2 | 23
  Any Solicited Local Reactogenicity Event: Moderate (Grade 2) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Any Solicited Local Reactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Local Reactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: None | 8 | 12 | 10 | 9 | 12 | 14 | 15 | 18 | 80
  Pain/Tenderness: Mild (Grade 1) | 6 | 2 | 6 | 4 | 3 | 1 | 0 | 2 | 22
  Pain/Tenderness: Moderate (Grade 2) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Pain/Tenderness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Itching: None | 12 | 14 | 15 | 14 | 15 | 15 | 15 | 19 | 100
  Itching: Mild (Grade 1) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4
  Itching: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Itching: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Itching: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: None | 14 | 14 | 15 | 13 | 14 | 15 | 15 | 20 | 100
  Warmth: Mild (Grade 1) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 4
  Warmth: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: None | 13 | 14 | 15 | 14 | 15 | 15 | 15 | 20 | 101
  Swelling/Induration: Mild (Grade 1) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Swelling/Induration: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: None | 14 | 14 | 16 | 14 | 14 | 15 | 15 | 20 | 102
  Redness/Erythema: Mild (Grade 1) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Redness/Erythema: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: None | 15 | 14 | 16 | 14 | 15 | 15 | 15 | 20 | 104
  Hardness: Mild (Grade 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Solicited Local Events Post Vaccination 5 by Vaccination Group (Outcome 5)
Description: Incidence (number and percentage of participants) of local reactogenicity events post dose 5 by symptom, maximum severity, and priming dose group
Time Frame: Day 1-Day 7 Post Vaccination 5
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 2: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel®/ ALF43 | Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel | Group 4: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 5: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 6: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 7: | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 12 | 14 | 13 | 15 | 14 | 15 | 14 | 21 | 97
Participants
  Any Solicited Local Reactogenicity Event: None | 10 | 12 | 11 | 13 | 12 | 14 | 14 | 20 | 86
  Any Solicited Local Reactogenicity Event: Mild (Grade 1) | 2 | 2 | 2 | 2 | 2 | 1 | 0 | 1 | 11
  Any Solicited Local Reactogenicity Event: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Local Reactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Local Reactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: None | 10 | 12 | 11 | 14 | 12 | 14 | 14 | 20 | 87
  Pain/Tenderness: Mild (Grade 1) | 2 | 2 | 2 | 1 | 2 | 1 | 0 | 1 | 10
  Pain/Tenderness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Itching: None | 11 | 14 | 13 | 15 | 14 | 15 | 14 | 21 | 96
  Itching: Mild (Grade 1) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Itching: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Itching: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Itching: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: None | 12 | 14 | 13 | 14 | 14 | 15 | 14 | 21 | 96
  Warmth: Mild (Grade 1) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Warmth: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: None | 12 | 14 | 12 | 15 | 14 | 15 | 14 | 21 | 96
  Swelling/Induration: Mild (Grade 1) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Swelling/Induration: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: None | 12 | 14 | 13 | 15 | 13 | 15 | 14 | 21 | 96
  Redness/Erythema: Mild (Grade 1) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Redness/Erythema: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: None | 11 | 14 | 13 | 15 | 14 | 15 | 14 | 21 | 96
  Hardness: Mild (Grade 1) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hardness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Solicited Local Events Post Vaccination 6 by Vaccination Group (Outcome 6)
Description: Incidence (number and percentage of participants) of local reactogenicity events post dose 6 by symptom, maximum severity, and vaccination group
Time Frame: Day 1-Day 7 Post Vaccination 6
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 2: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel®/ ALF43 | Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel | Group 4: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 5: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 6: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 7: | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 12 | 14 | 12 | 15 | 15 | 15 | 14 | 20 | 97
Participants
  Any Solicited Local Reactogenicity Event: None | 9 | 13 | 11 | 13 | 14 | 14 | 14 | 20 | 88
  Any Solicited Local Reactogenicity Event: Mild (Grade 1) | 3 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 9
  Any Solicited Local Reactogenicity Event: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Local Reactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Local Reactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: None | 11 | 13 | 11 | 13 | 14 | 15 | 14 | 20 | 91
  Pain/Tenderness: Mild (Grade 1) | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 6
  Pain/Tenderness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Itching: None | 10 | 14 | 12 | 15 | 15 | 14 | 14 | 20 | 94
  Itching: Mild (Grade 1) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Itching: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Itching: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Itching: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: None | 11 | 14 | 12 | 15 | 15 | 14 | 14 | 20 | 95
  Warmth: Mild (Grade 1) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Warmth: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Warmth: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: None | 11 | 14 | 12 | 14 | 15 | 15 | 14 | 20 | 95
  Swelling/Induration: Mild (Grade 1) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Swelling/Induration: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling/Induration: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: None | 12 | 14 | 12 | 15 | 15 | 15 | 14 | 20 | 97
  Redness/Erythema: Mild (Grade 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness/Erythema: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: None | 12 | 14 | 12 | 14 | 15 | 15 | 14 | 20 | 96
  Hardness: Mild (Grade 1) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Hardness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hardness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Solicited Systemic Events Post Vaccination 1 by Priming Dose Group (Outcome 7)
Description: Incidence (number and percentage of participants) of systemic reactogenicity events post dose 1 by symptom, maximum severity, and priming dose group
Time Frame: Day 1-Day 7 Post Vaccination 1
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Priming Dose Group 1: Prime of Env-C Plasmid DNA Alone | Priming Dose Group 2: Prime of Env-C Plasmid DNA / dmLT | Priming Dose Group 3: Prime of Env-C Plasmid DNA / ALF43 | Priming Dose Group 4: Prime of Env-C Plasmid DNA / ALF43 / HIV Env gp145 C.6980 Protein | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 33 | 32 | 33 | 16 | 23 | 114
Participants
  Any Solicited Systemic Reactogenicity Event: None | 17 | 21 | 16 | 8 | 12 | 62
  Any Solicited Systemic Reactogenicity Event: Mild (Grade 1) | 14 | 10 | 17 | 6 | 11 | 47
  Any Solicited Systemic Reactogenicity Event: Moderate (Grade 2) | 2 | 1 | 0 | 2 | 0 | 5
  Any Solicited Systemic Reactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Systemic Reactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Fever: number analyzed (Participants) | 33 | 32 | 33 | 16 | 22 | 114
  Fever: None | 31 | 31 | 33 | 13 | 21 | 108
  Fever: Mild (Grade 1) | 1 | 1 | 0 | 1 | 1 | 3
  Fever: Moderate (Grade 2) | 1 | 0 | 0 | 2 | 0 | 3
  Fever: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Fever: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: None | 21 | 26 | 26 | 11 | 17 | 84
  Fatigue/Tiredness: Mild (Grade 1) | 11 | 6 | 7 | 5 | 6 | 29
  Fatigue/Tiredness: Moderate (Grade 2) | 1 | 0 | 0 | 0 | 0 | 1
  Fatigue/Tiredness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 28 | 29 | 32 | 14 | 20 | 103
  Myalgia: Mild (Grade 1) | 4 | 3 | 1 | 2 | 3 | 10
  Myalgia: Moderate (Grade 2) | 1 | 0 | 0 | 0 | 0 | 1
  Myalgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 30 | 27 | 31 | 14 | 20 | 102
  Arthralgia: Mild (Grade 1) | 3 | 4 | 2 | 2 | 3 | 11
  Arthralgia: Moderate (Grade 2) | 0 | 1 | 0 | 0 | 0 | 1
  Arthralgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 19 | 23 | 20 | 11 | 12 | 73
  Headache: Mild (Grade 1) | 13 | 8 | 13 | 5 | 11 | 39
  Headache: Moderate (Grade 2) | 1 | 1 | 0 | 0 | 0 | 2
  Headache: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 29 | 27 | 32 | 14 | 20 | 102
  Chills: Mild (Grade 1) | 4 | 4 | 1 | 2 | 3 | 11
  Chills: Moderate (Grade 2) | 0 | 1 | 0 | 0 | 0 | 1
  Chills: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Rash: None | 33 | 32 | 32 | 16 | 23 | 113
  Rash: Mild (Grade 1) | 0 | 0 | 1 | 0 | 0 | 1
  Rash: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 32 | 31 | 32 | 13 | 21 | 108
  Nausea: Mild (Grade 1) | 1 | 1 | 1 | 3 | 2 | 6
  Nausea: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: None | 27 | 27 | 30 | 13 | 20 | 97
  Dizziness: Mild (Grade 1) | 5 | 5 | 3 | 3 | 3 | 16
  Dizziness: Moderate (Grade 2) | 1 | 0 | 0 | 0 | 0 | 1
  Dizziness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Solicited Systemic Events Post Vaccination 2 by Priming Dose Group (Outcome 8)
Description: Incidence (number and percentage of participants) of systemic reactogenicity events post dose 2 by symptom, maximum severity, and priming dose group
Time Frame: Day 1-Day 7 Post Vaccination 2
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Priming Dose Group 1: Prime of Env-C Plasmid DNA Alone | Priming Dose Group 2: Prime of Env-C Plasmid DNA / dmLT | Priming Dose Group 3: Prime of Env-C Plasmid DNA / ALF43 | Priming Dose Group 4: Prime of Env-C Plasmid DNA / ALF43 / HIV Env gp145 C.6980 Protein | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 30 | 25 | 31 | 15 | 20 | 101
Participants
  Any Solicited Systemic Reactogenicity Event: None | 22 | 17 | 25 | 9 | 15 | 73
  Any Solicited Systemic Reactogenicity Event: Mild (Grade 1)8 | 8 | 6 | 6 | 6 | 5 | 26
  Any Solicited Systemic Reactogenicity Event: Moderate (Grade 2 | 0 | 2 | 0 | 0 | 0 | 2
  Any Solicited Systemic Reactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Systemic Reactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Fever: None | 30 | 24 | 28 | 12 | 20 | 94
  Fever: Mild (Grade 1)8 | 0 | 0 | 3 | 3 | 0 | 6
  Fever: Moderate (Grade 2 | 0 | 1 | 0 | 0 | 0 | 1
  Fever: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Fever: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: None | 27 | 22 | 30 | 13 | 17 | 92
  Fatigue/Tiredness: Mild (Grade 1)8 | 3 | 3 | 1 | 2 | 3 | 9
  Fatigue/Tiredness: Moderate (Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 29 | 21 | 31 | 14 | 19 | 95
  Myalgia: Mild (Grade 1)8 | 1 | 4 | 0 | 1 | 1 | 6
  Myalgia: Moderate (Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 28 | 23 | 31 | 14 | 19 | 96
  Arthralgia: Mild (Grade 1)8 | 2 | 2 | 0 | 1 | 1 | 5
  Arthralgia: Moderate (Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 28 | 22 | 30 | 14 | 19 | 94
  Chills: Mild (Grade 1)8 | 2 | 3 | 1 | 1 | 1 | 7
  Chills: Moderate (Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 22 | 21 | 30 | 13 | 17 | 86
  Headache: Mild (Grade 1)8 | 8 | 3 | 1 | 2 | 3 | 14
  Headache: Moderate (Grade 2 | 0 | 1 | 0 | 0 | 0 | 1
  Headache: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Rash: None | 29 | 24 | 31 | 14 | 20 | 98
  Rash: Mild (Grade 1)8 | 1 | 1 | 0 | 1 | 0 | 3
  Rash: Moderate (Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 28 | 23 | 31 | 14 | 18 | 96
  Nausea: Mild (Grade 1)8 | 2 | 2 | 0 | 1 | 2 | 5
  Nausea: Moderate (Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: None | 27 | 23 | 30 | 14 | 20 | 94
  Dizziness: Mild (Grade 1)8 | 3 | 2 | 1 | 1 | 0 | 7
  Dizziness: Moderate (Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Solicited Systemic Events Post Vaccination 3 by Priming Dose Group (Outcome 9)
Description: Incidence (number and percentage of participants) of systemic reactogenicity events post dose 3 by symptom, maximum severity, and vaccination group
Time Frame: Day 1-Day 7 Post Vaccination 3
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Priming Dose Group 1: Prime of Env-C Plasmid DNA Alone | Priming Dose Group 2: Prime of Env-C Plasmid DNA / dmLT | Priming Dose Group 3: Prime of Env-C Plasmid DNA / ALF43 | Priming Dose Group 4: Prime of Env-C Plasmid DNA / ALF43 / HIV Env gp145 C.6980 Protein | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 30 | 24 | 30 | 14 | 20 | 98
Participants
  Any Solicited Systemic Reactogenicity Event: None | 20 | 21 | 26 | 12 | 18 | 79
  Any Solicited Systemic Reactogenicity Event: Mild (Grade 1) | 9 | 3 | 3 | 2 | 2 | 17
  Any Solicited Systemic Reactogenicity Event: Moderate (Grade 2) | 1 | 0 | 1 | 0 | 0 | 2
  Any Solicited Systemic Reactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Systemic Reactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Fever: None | 29 | 23 | 29 | 14 | 20 | 95
  Fever: Mild (Grade 1) | 0 | 1 | 0 | 0 | 0 | 1
  Fever: Moderate (Grade 2) | 1 | 0 | 1 | 0 | 0 | 2
  Fever: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Fever: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: None | 26 | 24 | 29 | 14 | 20 | 93
  Fatigue/Tiredness: Mild (Grade 1) | 4 | 0 | 1 | 0 | 0 | 5
  Fatigue/Tiredness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 29 | 24 | 29 | 14 | 20 | 96
  Arthralgia: Mild (Grade 1) | 1 | 0 | 1 | 0 | 0 | 2
  Arthralgia: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 29 | 24 | 29 | 13 | 20 | 95
  Myalgia: Mild (Grade 1) | 1 | 0 | 1 | 1 | 0 | 3
  Myalgia: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 22 | 22 | 28 | 12 | 18 | 84
  Headache: Mild (Grade 1) | 8 | 2 | 2 | 2 | 2 | 14
  Headache: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 28 | 24 | 30 | 13 | 19 | 95
  Chills: Mild (Grade 1) | 2 | 0 | 0 | 1 | 1 | 3
  Chills: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Rash: None | 30 | 24 | 30 | 14 | 20 | 98
  Rash: Mild (Grade 1) | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 29 | 24 | 29 | 14 | 20 | 96
  Nausea: Mild (Grade 1) | 1 | 0 | 1 | 0 | 0 | 2
  Nausea: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: None | 28 | 24 | 29 | 14 | 20 | 95
  Dizziness: Mild (Grade 1) | 2 | 0 | 1 | 0 | 0 | 3
  Dizziness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Solicited Systemic Events Post Vaccination 4 by Vaccination Group (Outcome 10)
Description: Incidence (number and percentage of participants) of systemic reactogenicity events post dose 4 by symptom, maximum severity, and vaccination group
Time Frame: Day 1-Day 7 Post Vaccination 4
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 2: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel®/ ALF43 | Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel | Group 4: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 5: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 6: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 7: | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 15 | 14 | 16 | 14 | 15 | 15 | 15 | 20 | 104
Participants
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: None | 8 | 11 | 12 | 10 | 13 | 12 | 13 | 16 | 79
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Mild (Grade 1) | 7 | 3 | 4 | 2 | 2 | 2 | 1 | 4 | 21
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Moderate (Grade 2) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 4
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fever: number analyzed (Participants) | 14 | 14 | 16 | 14 | 15 | 15 | 15 | 20 | 103
  Fever: None | 12 | 14 | 16 | 11 | 14 | 14 | 13 | 20 | 94
  Fever: Mild (Grade 1) | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 5
  Fever: Moderate (Grade 2) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 4
  Fever: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fever: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: None | 14 | 13 | 16 | 13 | 15 | 15 | 15 | 19 | 101
  Fatigue/Tiredness: Mild (Grade 1) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3
  Fatigue/Tiredness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 13 | 14 | 15 | 13 | 14 | 15 | 15 | 20 | 99
  Myalgia: Mild (Grade 1) | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 5
  Myalgia: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 15 | 14 | 15 | 14 | 15 | 14 | 15 | 19 | 102
  Arthralgia: Mild (Grade 1) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2
  Arthralgia: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 10 | 12 | 12 | 12 | 15 | 14 | 15 | 16 | 90
  Headache: Mild (Grade 1) | 5 | 2 | 4 | 2 | 0 | 1 | 0 | 4 | 14
  Headache: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 15 | 13 | 16 | 12 | 14 | 15 | 15 | 20 | 100
  Chills: Mild (Grade 1) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 4
  Chills: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: None | 15 | 14 | 16 | 14 | 15 | 15 | 15 | 20 | 104
  Rash: Mild (Grade 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 14 | 13 | 16 | 14 | 15 | 15 | 15 | 20 | 102
  Nausea: Mild (Grade 1) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Nausea: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: None | 13 | 14 | 15 | 14 | 15 | 15 | 15 | 20 | 101
  Dizziness: Mild (Grade 1) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Dizziness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Solicited Systemic Events Post Vaccination 5 by Vaccination Group (Outcome 11)
Description: Incidence (number and percentage of participants) of systemic reactogenicity events post dose 5 by symptom, maximum severity, and priming dose group
Time Frame: Day 1-Day 7 Post Vaccination 5
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 2: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel®/ ALF43 | Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel | Group 4: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 5: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 6: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 7: | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 12 | 14 | 13 | 15 | 14 | 15 | 14 | 21 | 97
Participants
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: None | 8 | 9 | 12 | 14 | 14 | 13 | 12 | 16 | 82
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Mild (Grade 1) | 4 | 4 | 1 | 1 | 0 | 1 | 2 | 5 | 13
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Moderate (Grade 2) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fever: None | 10 | 14 | 13 | 15 | 14 | 14 | 13 | 17 | 93
  Fever: Mild (Grade 1) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3
  Fever: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Fever: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fever: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: None | 10 | 11 | 13 | 15 | 14 | 14 | 14 | 20 | 91
  Fatigue/Tiredness: Mild (Grade 1) | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 6
  Fatigue/Tiredness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 11 | 13 | 13 | 14 | 14 | 14 | 14 | 21 | 93
  Myalgia: Mild (Grade 1) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 4
  Myalgia: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 12 | 14 | 13 | 14 | 14 | 15 | 14 | 20 | 96
  Arthralgia: Mild (Grade 1) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Arthralgia: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 8 | 11 | 12 | 14 | 14 | 15 | 13 | 19 | 87
  Headache: Mild (Grade 1) | 4 | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 9
  Headache: Moderate (Grade 2) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Headache: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 11 | 12 | 13 | 14 | 14 | 15 | 14 | 21 | 93
  Chills: Mild (Grade 1) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 4
  Chills: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: None | 12 | 14 | 13 | 15 | 14 | 15 | 14 | 21 | 97
  Rash: Mild (Grade 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 11 | 13 | 12 | 14 | 14 | 15 | 14 | 21 | 93
  Nausea: Mild (Grade 1) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 4
  Nausea: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: None | 11 | 10 | 13 | 14 | 14 | 15 | 14 | 21 | 91
  Dizziness: Mild (Grade 1) | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 6
  Dizziness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Solicited Systemic Events Post Vaccination 6 by Vaccination Group (Outcome 12)
Description: Incidence (number and percentage of participants) of systemic reactogenicity events post dose 6 by symptom, maximum severity, and vaccination group
Time Frame: Day 1-Day 7 Post Vaccination 6
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 2: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel®/ ALF43 | Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel | Group 4: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 5: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 6: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Group 7: | Pooled Placebo | All Participants Receiving Env-C Plasmid DNA
Number analyzed (Participants) | 12 | 14 | 12 | 15 | 15 | 15 | 14 | 20 | 97
Participants
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: None | 8 | 12 | 9 | 12 | 11 | 14 | 13 | 16 | 79
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Mild (Grade 1) | 3 | 2 | 3 | 2 | 4 | 1 | 0 | 4 | 15
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Moderate (Grade 2) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Solicited Systemic Reactogenicity EventReactogenicity Event: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fever: None | 10 | 13 | 12 | 14 | 14 | 15 | 13 | 20 | 91
  Fever: Mild (Grade 1) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Fever: Moderate (Grade 2) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Fever: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fever: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: None | 12 | 14 | 11 | 15 | 15 | 14 | 14 | 18 | 95
  Fatigue/Tiredness: Mild (Grade 1) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2
  Fatigue/Tiredness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue/Tiredness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 12 | 14 | 10 | 15 | 13 | 15 | 14 | 20 | 93
  Myalgia: Mild (Grade 1) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 4
  Myalgia: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 12 | 14 | 11 | 15 | 14 | 15 | 14 | 20 | 95
  Arthralgia: Mild (Grade 1) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Arthralgia: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 11 | 13 | 9 | 14 | 14 | 14 | 14 | 17 | 89
  Headache: Mild (Grade 1) | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 3 | 8
  Headache: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 11 | 14 | 10 | 15 | 14 | 15 | 14 | 20 | 93
  Chills: Mild (Grade 1) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 4
  Chills: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: None | 12 | 14 | 12 | 15 | 15 | 15 | 14 | 20 | 97
  Rash: Mild (Grade 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 12 | 13 | 12 | 15 | 14 | 14 | 14 | 20 | 94
  Nausea: Mild (Grade 1) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3
  Nausea: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: None | 12 | 14 | 10 | 14 | 15 | 15 | 14 | 20 | 94
  Dizziness: Mild (Grade 1) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3
  Dizziness: Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness: Potentially Life-Threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Related Unsolicited AEs (Outcome 13)
Description: Incidence (number and percentage of participants) of related unsolicited AEs by maximum severity and vaccination group.
Time Frame: Day 1-Day 728
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel: Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 protein / Rehydragel
- Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel®: Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 protein / Rehydragel®
- Priming Dose Group 4: Prime of Env-C Plasmid DNA / dmLT / HIV Env gp145 C.6980 Protein (Group 7): Priming Dose Group 4: Prime of Env-C Plasmid DNA / dmLT / HIV Env gp145 C.6980 protein (Group 7)
Arm/Group | Priming Dose Group 1: Prime of Env-C Plasmid DNA Alone | Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel | Group 2: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel®/ ALF43 | Priming Dose Group 2: Prime of Env-C Plasmid DNA / dmLT | Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 4: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Priming Dose Group 3: Prime of Env-C Plasmid DNA / ALF43 | Group 5: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 6: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Priming Dose Group 4: Prime of Env-C Plasmid DNA / dmLT / HIV Env gp145 C.6980 Protein (Group 7) | Pooled Placebo
Number analyzed (Participants) | 33 | 17 | 16 | 32 | 16 | 16 | 33 | 16 | 17 | 16 | 23
Participants
  Mild Grade 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Moderate / Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe / Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potentially Life-Threatening / Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  None | 32 | 16 | 16 | 32 | 16 | 16 | 32 | 15 | 17 | 16 | 23

14. Primary Outcome: Number of SAEs (Outcome 14)
Description: Incidence (number and percentage of participants) of SAEs by maximum severity and vaccination group
Time Frame: Day 1-Day 728
Population: The safety population includes all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Priming Dose Group 1: Prime of Env-C Plasmid DNA Alone | Group 1: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel | Group 2: Env-C Plasmid DNA + HIV Env gp145 C.6980 Protein / Rehydragel®/ ALF43 | Priming Dose Group 2: Prime of Env-C Plasmid DNA / dmLT | Group 3: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 4: Env-C Plasmid DNA + dmLT + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Priming Dose Group 3: Prime of Env-C Plasmid DNA / ALF43 | Group 5: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® | Group 6: Env-C Plasmid DNA / ALF43 + HIV Env gp145 C.6980 Protein / Rehydragel® / ALF43 | Priming Dose Group 4: Prime of Env-C Plasmid DNA / dmLT / HIV Env gp145 C.6980 Protein (Group 7) | Pooled Placebo
Number analyzed (Participants) | 33 | 17 | 16 | 32 | 16 | 16 | 33 | 16 | 17 | 16 | 23
Participants
  Mild Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Moderate / Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe / Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potentially Life-Threatening / Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  None | 32 | 16 | 16 | 32 | 16 | 16 | 33 | 16 | 17 | 16 | 23

15. Secondary Outcome: Magnitude of Plasma IgG Binding Antibodies in Response to Differing DNA Priming Regimens
Description: Measured by binding antibody assays.
Time Frame: Thru Week 105
Reporting Status: Not Posted

16. Secondary Outcome: Durability of Plasma IgG Binding Antibodies in Response to Differing DNA Priming Regimens
Description: Measured by binding antibody assays.
Time Frame: Thru Week 105
Reporting Status: Not Posted

17. Secondary Outcome: Area Under the Curve (AUC) for Plasma IgG Binding Antibodies in Response to Differing DNA Priming Regimens
Description: Measured by binding antibody assays.
Time Frame: Thru Week 105
Reporting Status: Not Posted

18. Secondary Outcome: Magnitude of Plasma IgG Binding Antibodies Between Groups With and Without Rehydragel® After HIV Env gp145 C.6980 Protein Boosting
Description: Measured by binding antibody assays.
Time Frame: Thru Week 105
Reporting Status: Not Posted

19. Secondary Outcome: Durability of Plasma IgG Binding Antibodies Between Groups With and Without Rehydragel® After HIV Env gp145 C.6980 Protein Boosting
Description: Measured by binding antibody assays.
Time Frame: Thru Week 105
Reporting Status: Not Posted

20. Secondary Outcome: AUC for Plasma IgG Binding Antibodies Between Groups With and Without Rehydragel® After HIV Env gp145 C.6980 Protein Boosting
Description: Measured by binding antibody assays.
Time Frame: Thru Week 105
Reporting Status: Not Posted

21. Secondary Outcome: Presence of Plasma IgG Binding Antibodies
Description: Functional antibodies assessed using rapid fluorometric Antibody-dependent Cell-Mediated Cytotoxicity (ADCC) Assay, Antibody-dependent Cell-mediated Phagocytosis (ADCP), Antibody-dependent Complement (ADC) activation assays, or other functional assays. Neutralizing antibodies assessed using cell line-based and PBMC assays with a panel of viruses from different HIV subtypes, including A, B, C, D, and other circulating recombinant forms (CRFs) such as AE and AG.
Time Frame: Thru Week 105
Reporting Status: Not Posted

22. Secondary Outcome: Presence of Plasma IgA Binding Antibodies
Description: as for outcome 21
Time Frame: Thru Week 105
Reporting Status: Not Posted

23. Secondary Outcome: Types of Cell-mediated Immune Responses
Description: Cryopreserved PBMC and lymph nodes will be stimulated with HIV-1-specific antigens and tested using standard (but not limited to) cellular immune assays which may include but are not limited to Intracellular cytokine Staining, ELISPOT, Lymphoproliferation assays, B-cell analysis, T-follicular helper cell and innate immune cell analysis.
Time Frame: Thru Week 105
Reporting Status: Not Posted

24. Secondary Outcome: Level of Cell-mediated Immune Responses
Description: as for outcome 23
Time Frame: Thru Week 105
Reporting Status: Not Posted

25. Secondary Outcome: Types of Mucosal Humoral Responses
Description: Including, but not limited to, plasma IgG and IgA binding antibodies to HIV Env proteins, IgG and IgA subclass, and functional assays.
Time Frame: Thru Week 104
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs will be assessed and followed from initial recognition of the AE through end of the protocol defined follow-up period. SAEs will be followed up through resolution even if duration of followup goes beyond the protocol-defined the follow-up period. Adverse Events will be followed through the end of the study, a full 12 months following the last vaccination.
Description: ICH E6 defines an AE as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. FDA defines an AE as any untoward medical occurrence associated with the use of a drug in humans, whether considered drug related.
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Group 7: Vaccine | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 0/16 | 0/16 | 0/16 | 0/17 | 0/16 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/16 | 0/16 | 0/16 | 0/16 | 0/17 | 0/16 | 0/23
Other Adverse Events (participants affected / at risk) | 15/17 | 15/16 | 14/16 | 13/16 | 13/16 | 13/17 | 13/16 | 17/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=17) | Group 2: Vaccine (N=16) | Group 3: Vaccine (N=16) | Group 4: Vaccine (N=16) | Group 5: Vaccine (N=16) | Group 6: Vaccine (N=17) | Group 7: Vaccine (N=16) | Pooled Placebo (N=23)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Type 1 diabetes mellitus
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=17) | Group 2: Vaccine (N=16) | Group 3: Vaccine (N=16) | Group 4: Vaccine (N=16) | Group 5: Vaccine (N=16) | Group 6: Vaccine (N=17) | Group 7: Vaccine (N=16) | Pooled Placebo (N=23)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 3 (5) | 1 (1)
Leukopenias NEC (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graves' disease (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amoebiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrapulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 3 (3) | 6 (6) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 10 (12) | 4 (6) | 6 (9) | 5 (6) | 4 (5) | 4 (6) | 3 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 3 (3)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wound infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 3 (4) | 1 (1) | 5 (5) | 4 (4)
International normalised ratio increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 6 (6) | 4 (6) | 3 (5) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT04826094/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT04826094/SAP_001.pdf